CLINICAL TRIAL: NCT00476866
Title: Intermittent Positive-Pressure Breathing Effects in Patients With High Spinal Cord Injury
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: The number of patients desired has been reached
Sponsor: University of Versailles (Other)
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: CIT-17
Record Dates: First submitted 2007-05-21; First posted 2007-05-22 (Estimated); Last update posted 2007-05-22 (Estimated); Status verified 2007-05

CONDITIONS: Central Cord Injury Syndrome; Central Spinal Cord Syndrome
Keywords: Paraplegia; tetraplegia; lung compliance; work of breathing; hyperinflation; rehabilitation
MeSH Terms: conditions — Central Cord Syndrome; Paraplegia; Quadriplegia | interventions — Intermittent Positive-Pressure Breathing

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Device: intermittent positive-pressure breathing (IPPB)

SUMMARY:
Background: To determine whether intermittent positive-pressure breathing (IPPB) improved lung compliance, work of breathing, and respiratory function in patients with recent high spinal cord injury (SCI).

Methods: Two months of IPPB and two months of conventional treatment have to evaluated prospectively in random order in 14 patients with SCI. Noninvasive lung function tests and arterial blood gas measurements have to be obtained repeatedly. Repeated measurements of dynamic compliance and work of breathing have to be performed in 7 of the 14 patients.

DETAILED DESCRIPTION:
Patients The local ethics committee approved the study, and all patients have to give their written informed consent prior to inclusion. To be included patients had to satisfy the following criteria: (a) American Spinal Injury Association (ASIA) Class A or B10 SCI caused by trauma within the last 6 months and located between C5 and T6, (b) no thoracic injury, (c) and admission to a rehabilitation unit. The study was conducted over the first 4 months in the rehabilitation unit.

Measurements All tests will be performed with the patients seated in their wheelchairs. Lung function was tested using a Vmax 229 Sensormedics System (Yorba Linda, CA) according to standard guidelines.11 Arterial blood gas levels will be measured in capillary blood immediately after sampling from the radial artery with local anesthesia (topical lidocaine prilocaine, Emla®, Astra, Westborough, ME), using a Radiometer ABL 330 analyzer (Tacussel Radiometer Analytical, Copenhagen, Denmark). Flow will be measured using a Fleisch #2 pneumotachograph (Lausanne, Switzerland) and esophageal pressure (Pes) using a catheter-mounted pressure transducer system (Gaeltec, Dunvegan, UK). Appropriate placement will be verified by the occlusion test.12

Data Analysis Respiratory parameters will bemeasured during the last 5 minutes of a 20-minute period of relaxed breathing. From the flow tracings, we will measure inspiratory time (TI) and respiratory frequency (fR). Tidal volume (VT) will be obtained from the integrated flow signal. Dynamic lung compliance (CLdyn) will be calculated as the ratio of VT over the Pes difference at the points of zero flow corresponding to the start and end of inspiration.13 Inspiratory WOB (joule/min) will be calculated from a Campbell diagram by computing the area enclosed between the inspiratory Pes-VT curve and the theoretical static pressure-volume curve of the chest wall, as previously described.14 In addition, WOB will be partitioned into its elastic (WOBel) and resistive (WOBres) components on either side of the line joining the two zero-flow points.

Study protocol All patients will be studied during 2 months with and 2 months without IPPB, in random order. IPPB treatment will consist in at least 20 minutes of IPPB twice a day and 5 days a week. The patient will be comfortably seated with the back of the chair inclined at 45°. Inspiratory pressure will increase gradually to either the highest tolerated value or 40 cm H2O. Respiratory rate, inspiratory flow (from 20 to 60 L/min), and end-inspiratory trigger will be set to maximize patient comfort. The patients chose between a mouthpiece (Bird, Palm Springs, CA) and a nasal mask (Respironics, Herrsching, Germany). During both of the 2-month treatment periods, the number of patients who will require physiotherapy to clear excess secretions and the number of physiotherapy sessions per patient will be recorded.

Lung function tests will be performed at inclusion and at the end of each 2-month period in all patients. In addition, patients will be asked whether they will agree to measurements of flow, Pes, and gastric pressure at inclusion and at the end of each period. Measurements at the end of the IPPB period will be performed twice, immediately before and immediately after 20 minutes of IPPB with the catheter-mounted pressure-transducer system still in place. Each measurement period wil last about 5 minutes.

STATISTICS All data will be given as means±SD. Paired t tests will be used for within-patient comparisons of variables between the two treatments

ELIGIBILITY:
Inclusion Criteria:

* American Spinal Injury Association (ASIA) Class A or B10
* SCI caused by trauma within the last 6 months and located between C5 and T6
* admission to a rehabilitation unit.

Exclusion Criteria:

* thoracic injury

Min Age: 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 14 (Actual)
Dates: Start 2002-12; Study Completion 2005-03 (Actual)

PRIMARY OUTCOMES:
Vital capacity, lung compliance and work of breathing | 30 minutes after 2b months of treatment

SECONDARY OUTCOMES:
pulmonary function and blood gaz sample | 30 minutes after 2 months of treatment

CONTACTS AND LOCATIONS:
Overall Officials: Frédéric Lofaso, MD PhD, Principal Investigator — Assistance Publique-Hôpitaux de Paris and University of Versailles
Locations (1):
- Innovation Technological Center-Hôpital R. Poincaré, Garches, France

REFERENCES:
- [Background] McCool FD, Mayewski RF, Shayne DS, Gibson CJ, Griggs RC, Hyde RW. Intermittent positive pressure breathing in patients with respiratory muscle weakness. Alterations in total respiratory system compliance. Chest. 1986 Oct;90(4):546-52. doi: 10.1378/chest.90.4.546. PMID 3530648
- [Background] Trebbia G, Lacombe M, Fermanian C, Falaize L, Lejaille M, Louis A, Devaux C, Raphael JC, Lofaso F. Cough determinants in patients with neuromuscular disease. Respir Physiol Neurobiol. 2005 Apr 15;146(2-3):291-300. doi: 10.1016/j.resp.2005.01.001. PMID 15766917
- [Derived] Laffont I, Bensmail D, Lortat-Jacob S, Falaize L, Hutin C, Le Bomin E, Ruquet M, Denys P, Lofaso F. Intermittent positive-pressure breathing effects in patients with high spinal cord injury. Arch Phys Med Rehabil. 2008 Aug;89(8):1575-9. doi: 10.1016/j.apmr.2007.12.037. Epub 2008 Jul 7. PMID 18602082